CLINICAL TRIAL: NCT03551028
Title: Cultural Acceptability and Feasibility of HPV Cervical Self Collection Aided by the Mobile
Brief Title: HPV DNA Testing Through Mobile Mammography Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Emma McKim Mitchell, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19110
Record Dates: First submitted 2017-05-01; First posted 2018-06-11 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HPV self collection (Other): Pairing self-collection of HPV samples for DNA testing with women seeking mobile mammography.
  Interventions: Device: HPV self collection

INTERVENTIONS:
Device: HPV self collection — The proposed community based participatory study aims to determine whether offering self-collection for HPV testing through the mobile mammography unit is an acceptable and feasible method to increase access to cervical cancer screening for under-screened women in Southwest Virginia.

SUMMARY:
Invasive cervical cancer incidence and mortality can be dramatically reduced through early detection and treatment, but many women do not complete screening at recommended intervals. Many low-income women in Virginia remain uninsured and are at significant risk of being medically underserved and failing to complete regular cervical cancer screening. Self-collection of specimens for HPV testing is an innovative approach that may increase access to cervical cancer screening in populations that do not participate in traditional clinic-based screening. Innovative delivery models are needed to reach at-risk populations. This study seeks to explore the acceptability and feasibility of pairing self-collection of HPV samples for DNA testing with mobile mammography in women living in rural Virginia.

DETAILED DESCRIPTION:
The proposed study aims to determine whether offering self-collection for HPV testing through the mobile mammography unit is an acceptable and feasible method to increase access to cervical cancer screening for under-screened women in rural Virginia. The procedures will be recruitment of under-screened women in rural Virginia to complete HPV testing using self-collection kits distributed through the mobile mammography unit. Regardless of HPV positivity, all women will be provided with information about cervical cancer screening (locations, cost, etc.), and will be encouraged to complete Pap screening by a clinician.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant

Exclusion Criteria:

* history of hysterectomy or pelvic RT non English speaking

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Mitchell, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gravitt PE, Belinson JL, Salmeron J, Shah KV. Looking ahead: a case for human papillomavirus testing of self-sampled vaginal specimens as a cervical cancer screening strategy. Int J Cancer. 2011 Aug 1;129(3):517-27. doi: 10.1002/ijc.25974. PMID 21384341
- [Background] Balasubramanian A, Kulasingam SL, Baer A, Hughes JP, Myers ER, Mao C, Kiviat NB, Koutsky LA. Accuracy and cost-effectiveness of cervical cancer screening by high-risk human papillomavirus DNA testing of self-collected vaginal samples. J Low Genit Tract Dis. 2010 Jul;14(3):185-95. doi: 10.1097/LGT.0b013e3181cd6d36. PMID 20592553

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV Self Collection
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who were due for breast and cervical screening, seeking mobile mammography
Arm/Group | HPV Self Collection
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Self-Collection Paired With Mobile Mammography
Description: Assess the cultural acceptability of self-collection for HPV testing among under-screened women in Southwest Virginia specifically who were seeking a mammogram at an episodic clinic. The outcome measure of ACCEPTABILITY was measured through: participants who opted in, or uptake of HPV self collection (yes/no); and intention to follow up upon learning of result.
Time Frame: 1 month (to allow for time to process samples and communicate results)
Population: Participants seeking mobile mammography at an episodic clinic in far Southwest Virginia (Planning Districts 1 and 2) were screened for eligibility and recruited for this study. Acceptability was measured by participant's uptake of self-collection (y/n). Of the 33 participants, 100% participated in self-collection of samples for HPV testing.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Self Collection
Number analyzed (Participants) | 33
Participants | 33

2. Primary Outcome: Feasibility of Self-Collection for HPV Paired With Mobile Mammography
Description: Assess the feasibility of self-collection for HPV testing among under-screened women in Southwest Virginia who were seeking a mammogram at an episodic clinic. FEASIBILITY was measured through: participant uptake of HPV self collection (yes/no); observations of clinic flow (i.e. how did this additional screening fit in with existing mammography services); and quality of samples collected (were any collected inaccurately or in a way that was impossible to detect).
Time Frame: 1 month (to allow for time to process samples and communicate results)
Population: Participants seeking mobile mammography at an episodic clinic in far Southwest Virginia (Planning Districts 1 and 2) were screened for eligibility and recruited for this study. Feasibility was measured by participant's uptake of self-collection (y/n) and quality of samples collected for testing. Of the 33 participants, 100% of samples collected yielded results.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Self Collection
Number analyzed (Participants) | 33
Participants | 33

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | HPV Self Collection
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03551028/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03551028/ICF_001.pdf